CLINICAL TRIAL: NCT05049083
Title: A Single-centre, Single-dose, Random, Open, Two-period, Cross-over Relative Bioavailability Study of Different Processes of SHR2554 Tablets in Healthy Adult Subjects
Brief Title: A Relative Bioavailability Study of Different Processes of SHR2554 Tablets in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SHR2554-I-108
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Intervention Model Description: A single-centre, single-dose, random, open, two-period, cross-over relative bioavailability study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: New Process SHR2554 tablet、Former Process SHR2554 tablet
- Treatment group B (Experimental)
  Interventions: Drug: Former Process SHR2554 tablet、New Process SHR2554 tablet

INTERVENTIONS:
Drug: New Process SHR2554 tablet、Former Process SHR2554 tablet — New Process, 350 mg SHR2554 tablets on study day 1 - Former Process, 350 mg SHR2554 tablets on study day 8
  Arms: Treatment group A
Drug: Former Process SHR2554 tablet、New Process SHR2554 tablet — Former Process, 350 mg SHR2554 tablets on study day 1 - New Process, 350 mg SHR2554 tablets on study day 8
  Arms: Treatment group B

SUMMARY:
TThe study is being conducted to evaluate the relative bioavailability, pharmacokinetics and safety of different tablet processes of SHR2554 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent and willing and able to participate this research.
2. Health female or male aged 18 to 45 at date of informed consent.
3. Weighing ≥45 kg for female and ≥50 kg for male, body mass index between 19.0 and 26.0 kg/m2.
4. Normal or abnormal but with no clinically significant in physical examination, vital signs, laboratory tests (haematology, clinical chemistry, urinalysis, coagulation function), 12 lead ECG, abdominal B ultrasound and CT.
5. Participants should have no fertility plan and take effective contraceptive measures voluntarily from 2 weeks prior dose (for female) until 3 months after the last dose (for both female and male), and have no sperm or ovum donation plan; for fertile women the serum HCG test must be negative within Screening.

Exclusion Criteria:

1. Participants with chronic or serious disease history or current disease in respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, mental system, etc., and are not suitable for enrollment as assessed by the investigator.
2. Surgery history that may affect drug absorption in gastrointestinal tract (including gastrectomy, enterectomy, stomach reduction surgery, etc.).
3. Surgery history within 6 months prior to screening or surgery plans during the study.
4. Plasma donation or blood loss greater than 400 mL or transfusion within 3 months prior to screening, or greater than 200 mL within 1 month prior to screening.
5. Positive results on screening tests for HBsAg and/or HCsAg and/or HIV and/or syphilis.
6. History of drug abuse or positive results of drug tests.
7. Alcohol abuse or smokers (≥14 units of alcohol per week within 6 months prior to screening: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine; ≥5 cigarettes per day), or unable to stop drinking or smoking during the study; positive results on screening tests for alcohol or nicotine.
8. History of allergy/hypersensitivity (allergy/hypersensitivity to more than two substances), or are not suitable for enrollment as assessed by the investigator.
9. Swallowing resistance or obstacles that affect drug absorption.
10. Participation in any other clinical study that included drug treatment within 3 months prior to first SHR2554 dose.
11. Administration of any CYP3A4 inducers or inhibitors within 4 weeks prior to first SHR2554 dose.
12. Administration of any prescription/non-prescription medicine or traditional Chinese medicine or dietary supplement within 2 weeks prior to first SHR2554 dose.
13. Administration of food or drinks that containing grapefruit, methylxanthine or alcohol within 72 hours prior to first SHR2554 dose; Strenuous exercise.
14. Participants who have special dietary requirements and cannot accept a unified diet.
15. Any factors that affect drug absorption, distribution, metabolism or excretion.
16. Lactating women.
17. History of fainting needles or blood; difficulty in blood collection or intolerance of venipuncture blood collection.
18. Any factors are not suitable for enrollment as assessed by the investigator or participants withdrew from the study for their own reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-01-06 (Estimated); Study Completion 2022-04-29 (Estimated)

PRIMARY OUTCOMES:
Cmax | day 1 to day 11
AUC0-t | day 1 to day 11
AUC0-∞ | day 1 to day 11
Tmax | day 1 to day 11
t1/2 | day 1 to day 11
CL/F | day 1 to day 11
Vz/F | day 1 to day 11

SECONDARY OUTCOMES:
The incidence and severity of adverse events/serious adverse events | from ICF signing date to approximate day 15

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided